CLINICAL TRIAL: NCT02820181
Title: Assessment of Functionality and Performance of a Novel Tracheostomy Tie
Brief Title: Assessment of a Novel Tracheostomy Tie
Acronym: AONTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Jun Tian, Associate Professor, The First Affiliated Hospital of Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FirstTianjunENT
Record Dates: First submitted 2016-06-22; First posted 2016-06-30 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Tracheostomy Complication
Keywords: tracheostomy ties

ARMS (2):
- novel tracheostomy bi-ties (Experimental): those with the novel tracheostomy bi-ties
  Interventions: Device: novel tracheostomy bi-ties
- traditional tracheostomy tie (Active Comparator): those with traditional tracheostomy tie
  Interventions: Device: traditional Tracheostomy ties

INTERVENTIONS:
Device: novel tracheostomy bi-ties — The investigators designed a novel tracheostomy bi-tie to ensure the safety and conveniences during exchanging and cleaning them, the primary feature of which is double belts and easy to operate.
  Arms: novel tracheostomy bi-ties
Device: traditional Tracheostomy ties — Traditionally, the tracheostomy tube is fixed using ordinary tracheostomy ties made of medical bandage or long strands.
  Arms: traditional tracheostomy tie

SUMMARY:
Tracheotomy is a common procedure for multiple medical indications.Tracheostomy tubes must be securely fixed to prevent movement or decannulation and tracheostomy ties must be exchanged as needed. However, the process of ties exchange is always risky and complicated. A novel tracheostomy tie has been designed to ensure the safety during exchanging and conveniences of cleaning. This study is to determine if the new device is better than the old one.

DETAILED DESCRIPTION:
Tracheotomy is a common procedure for multiple medical indications. Nursing staff must understand the immediate postoperative and long-term management of tracheostomy patients. To provide safe and competent care, tracheostomy tubes must be taken care of carefully, including cleaning or changing the inner cannula, caring for the stoma, suctioning at least 3 times a day, and replacing tracheostomy ties according to facility-specific policy as needed. However, to avoid inadvertent dislodgement of the tracheostomy tube, the process of ties exchange is always risky and complicated, which request one person to hold the tube in place while a second person performs the tie exchange.

The investigators designed a novel tracheostomy tie to ensure the safety during exchanging and conveniences of cleaning, the primary feature of which is double belts and easy to operate. This randomized controlled trial is to determine if the new device is better than the traditional one.

Sixty tracheotomy patients without an existing neck injury will be recruited . Patients in experimental group wear a novel tracheostomy tie. The traditional one was used in control group. Difficulty level of exchanging or cleaning the tracheostomy ties, degree of comfort, skin breakdown and the actually frequency of exchanging will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years old and ≤ 60 years old;
2. Patients with a tracheostomy;
3. With intact neck skin;
4. Willingly signs the Informed Consent;
5. Is qualified to participate in the opinion of the Investigator;
6. Without disorders of consciousness.

Exclusion Criteria:

1. With an existing neck injury or infection or clinically significant skin diseases on the application site which may contraindicate participation, including psoriasis, eczema, atopic dermatitis, active cancer;
2. With damaged skin or conditions on the application site which includes sunburn, scars, moles or other disfiguration of the test site;
3. Has a known or stated allergy to adhesive bandages, or any of the product types being tested;
4. Uses of topical drugs on the application site;
5. Uses lotions, creams or oils on the application site;
6. Can not communicate with nurses or doctors for any reasons

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binquan Wang, Study Director — The First Affiliated Hospital of Shanxi Medical University
Locations (1):
- The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Novel Tracheostomy Bi-ties | Traditional Tracheostomy Tie
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Novel Tracheostomy Bi-ties | Traditional Tracheostomy Tie | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (2.9) | 53.0 (5.5) | 53.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 28 | 29 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale to Measure the Difficulty Level of Exchanging or Cleaning the Tracheostomy Ties (0 to 10 ) Higher Scores Mean a Worse Outcome
Description: Nurses will be evaluated by Visual Analogue Scale/Score to measure the difficulty level of exchanging or cleaning the tracheostomy ties.
  Title: Visual Analogue Scale to measure the difficulty level of exchanging or cleaning the tracheostomy ties (0 to 10 ) Higher scores mean a worse outcome
Time Frame: 14days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Novel Tracheostomy Bi-ties | Traditional Tracheostomy Tie
Number analyzed (Participants) | 30 | 30
score on a scale | 1.2 (0.6) | 7.5 (0.5)

2. Primary Outcome: Number of Participants With Local Skin Breakdown
Description: Scale for breakdown of neck skin wound was rated as mild, moderate, or severe. "Mild" wounds included fragile skin that was erythematous or had a small amount of breakdown (<1 cm in diameter). Wounds with evident skin erosion or breakdown associated with drainage and/or pain were classified as "moderate." "Severe" wounds were defined as a partial-thickness loss of dermis presenting as a shallow open ulcer with a red-pink wound bed.
Time Frame: 14days
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Tracheostomy Bi-ties | Traditional Tracheostomy Tie
Number analyzed (Participants) | 30 | 30
Participants
  None | 30 | 27
  Mild | 0 | 2
  Moderate | 0 | 1
  Severe | 0 | 0

3. Secondary Outcome: Visual Analogue Scale of Comfort of Patients During Wearing or Exchanging Tracheostomy Ties (0-10) Higher Scores Mean Worse Outcome.
Description: Visual Analogue Scale/Score will be used to measure the degree of comfort of patients during wearing or exchanging tracheostomy ties Title: Visual Analogue Scale of comfort of patients during wearing or exchanging tracheostomy ties(0-10) Higher scores mean worse outcome.
Time Frame: 14days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Novel Tracheostomy Bi-ties | Traditional Tracheostomy Tie
Number analyzed (Participants) | 30 | 30
units on a scale | 1.0 (0.7) | 8.9 (0.8)

4. Secondary Outcome: Objective Index:the Actually Frequency of Exchanging Dressing
Description: The record of the frequency of exchanging dressing under the tracheostomy ties in practice will be collected
Time Frame: 14days
Measure: Mean (Standard Deviation); unit: Times
Arm/Group | Novel Tracheostomy Bi-ties | Traditional Tracheostomy Tie
Number analyzed (Participants) | 30 | 30
Times | 0 (0) | 2 (0.64)

ADVERSE EVENTS:
Time Frame: 14 days.
Arm/Group | Novel Tracheostomy Bi-ties | Traditional Tracheostomy Tie
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02820181/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02820181/ICF_001.pdf